CLINICAL TRIAL: NCT04772677
Title: Building Emotional Awareness and Mental Health - A Mobile App-Based Parenting Program for Depressed Mothers of Infants and Preschoolers, Matched With Unified Protocol Therapy Skills
Brief Title: Building Emotional Awareness and Mental Health
Acronym: BEAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: University of Calgary (Other); Tactica Interactive (Unknown); Centre for Healthcare Innovation (Unknown); Research Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEAM Pilot
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-02

CONDITIONS: Maternal Depression

STUDY DESIGN:
Intervention Model Description: This pilot study will include two arms. The first arm will enroll 30 mothers with children aged 6-17 months (i.e., infant cohort). The second arm will enroll 30 mothers with children aged 18-36 months (i.e., preschool cohort). The postpartum cohort will receive access to the online psychoeducation and social-connection platform and the preschool cohort will be randomized to the program or a services as usual control group. Analyses will be performed separately per each arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEAM - Infant (Experimental): BEAM Infant will be delivered via mobile application to mothers with a 6-17 month old child. It will include 15-30-minute lessons on mental health and parenting and a closed community forum. Mental Health videos will provide information and tools via The Unified Protocol, a best-practice program to address dysregulated emotions across mood and anxiety disorders. Parenting videos will help parents understand their children's challenging behaviours and teach proactive approaches to prevent negative interactions and promote a positive relationship. A closed online community forum will be facilitated by a mental health clinician and parent coach. Weekly Zoom meetings will be facilitated by clinicians where participants can meet with other participants, ask questions about the program content, or discuss the week's materials.
  Interventions: Behavioral: BEAM Mental Health and Parenting Program
- BEAM - Preschool (Experimental): BEAM Preschool will be delivered via mobile application to mothers with a 18-36 month old child. It will include 15-30-minute lessons on mental health and parenting and a closed community forum. Mental Health videos will provide information and tools via The Unified Protocol, a best-practice program to address dysregulated emotions across mood and anxiety disorders. Parenting Videos will help parents understand their children's challenging behaviours and teach proactive approaches to prevent negative interactions and promote a positive relationship. A closed online community forum will be facilitated by a mental health clinician and parent coach. Weekly Zoom meetings will be facilitated by clinicians where participants can meet with other participants, ask questions about the program content, or discuss the week's materials.
  Interventions: Behavioral: BEAM Mental Health and Parenting Program

INTERVENTIONS:
Behavioral: BEAM Mental Health and Parenting Program — The BEAM program is a novel mobile app-based therapeutic intervention that incorporates key parenting concepts and Unified Protocol (UP) therapy modules with clinician-facilitated peer social support and connection. The primary aim of the program is to improve symptoms of depression and promote a positive parent-child relationship. There are three main components of the program: 1) the UP content, which will target maternal mental health symptomology, 2) the parenting skills training content, which is designed to correspond to the UP modules and promote maternal responsivity to children's emotions, and 3) a closed online community forum to encourage social support and connection between participants of the program.

SUMMARY:
Since its emergence in December 2019, COVID-19 has reshaped the world. Mental health problems are predicted to rise dramatically as a secondary effect of the disease and measures put in place to contain it. Our emerging evidence shows parents of young children have not been spared from these effects and are experiencing 4-fold increases depression and anxiety. Young children are highly vulnerable to parent mental illness due to their reliance on caregivers to meet basic needs. Interventions are needed that consider the unique mental health and parenting challenges families are encountering during the pandemic. Our team of mental health and program development experts will address these needs through an online psychoeducation and social-connection platform, BEAM: Building Emotional Awareness and Mental Health. BEAM brings together best practices in online telehealth programs in a highly personalized and interactive format to address multiple family needs. With clinical research investigators across provinces, the BEAM pilot project will provide services to 60 mothers (30 per group) of 6-36 month old children in Manitoba and Alberta.

DETAILED DESCRIPTION:
Families are facing unprecedented challenges during the COVID-19 pandemic. Emerging evidence from our recent family research shows elevated rates of maternal depression in parents of 0-5-year-old children, compared to pre-pandemic cohorts with similar demographic profiles. In our combined data of over 3000 families of 0 to 5-year-old children, 37-48% of mothers were classified as depressed, based on child age group, with 65% of depressed mothers also experiencing anxiety. In early childhood, exposure to maternal mental illness predicts risk for children's own mental health problems, developmental delays, asthma, and injury risk. For mothers themselves, depression contributes to health problems and low quality of life. Notably, these harms are most pronounced when depression persists, highlighting the importance of intervening early to prevent intergenerational health impairments.

Although evidence-based treatments exist to address maternal mental illness, there are high barriers to accessing care due to COVID-19. These include physical distancing, high costs of individual therapy, closure of existing services, and overwhelming childcare demands. Only 5% of mothers in our sample with depression report accessing services in the past month. The parenting stress associated with maternal depression is established to lead to low-quality interactions and harsh discipline, which is particularly concerning with children are spending nearly all their time at home.

Addressing these intergenerational health concerns will require innovative program design methods to simultaneously treat maternal mental illness and address parenting risks. We have developed the Building Emotional Awareness & Mental Health (BEAM) program to immediately address these needs. Investing in maternal mental health now, before problems are entrenched, is expected to yield high health and economic benefits by preventing the long-term consequences of maternal depression from becoming embedded in children's biological and behavioural development. Our team of mental health, parenting, and program development experts will address these needs through an online psycho-education and social-connection platform.

There are 3 objectives for this study:

1. Support maternal mental wellness and parenting stress by creating an interactive psychoeducation & social connection online platform.
2. Evaluate the acceptability of the app and integrate parent feedback
3. Determine the potential benefits of BEAM on maternal and child well-being.

ELIGIBILITY:
Inclusion Criteria:

* Must have a 6-36 months old child
* Must have moderate-severe depression (i.e., a score of 10+ on the Patient Health Questionnaire)
* 18+ years of age
* comfortable understanding, speaking, and reading English
* Living in Manitoba or Alberta
* Must be available for weekly Zoom sessions

Exclusion Criteria:

* Child is outside the 6-36 month age range
* Lives outside of Manitoba or Alberta
* Does not meet criteria for moderate-severe depression
* A history of attempted suicide in past year or self-harm in past 6 months), or significant suicidal ideation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only mothers and other primary caregivers who identify as women (e.g., grandmothers, aunts) are eligible to participate.
Enrollment: 60 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Maternal Depression - Patient Health Questionnaire | PHQ-9 to be completed during eligibility screening, at T1 before starting the BEAM program, weekly for 10 weeks, at the end of the program (T2; 10 weeks), and at follow-up (T3; 18 weeks)
  Depression will be assessed with the Patient Health Questionnaire, a 9-item questionnaire will be used to measure depression presence and severity (mild to severe).
Change in Parenting Stress - Parent Daily Report | PDR to be completed at T1 before starting the BEAM Program, weekly for 10 weeks, at the end of the program (T2; 10 weeks), and at follow-up (T3; 18 weeks)
  Parenting stress will be assessed with the Parent Daily Report, a scale which contains 12 items assessing the presence of difficult child behaviours and whether they were stressful for parents.

SECONDARY OUTCOMES:
Change in Family Relationship Quality | To be assessed before starting the BEAM Program (T1), at the end of the program (T2; 10 weeks), and at follow-up (T3; 18 weeks)
  We will assess parent-child relationship quality and parenting strategies used by mothers through a collection of validated questionnaires (e.g., Parenting Stress Index, Parenting Scale), and the Couples Satisfaction Index will examine co-parent relationship quality in 2-parent households.
Change in Child and Family Function | To be assessed before starting the BEAM Program (T1), at the end of the program (T2; 10 weeks), and at follow-up (T3; 18 weeks)
  A variety of questionnaires will support the collection of data pertaining to child and family function, including other maternal mental health symptoms and psychological functioning(e.g., emotion regulation, anxiety, anger, self-compassion) , child mental health and behaviour (e.g., Child Behaviour Checklist), and the family environment (e.g., child and parent screen-time). All questionnaires are standardized and well-validated

OTHER OUTCOMES:
Change in Substance Use | To be assessed before starting the BEAM Program (T1), at the end of the program (T2; 10 weeks), and at follow-up (T3; 18 weeks)
  Mothers will be asked to report their use of alcohol, cannabis, tobacco and illicit drugs in the past month. In addition, the Alcohol Use Disorders Identification Test and a modified version of the Substance Use Motives Measure will be administered

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Manitoba - Department of Psychology, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Xie EB, Freeman M, Penner-Goeke L, Reynolds K, Lebel C, Giesbrecht GF, Rioux C, MacKinnon A, Sauer-Zavala S, Roos LE, Tomfohr-Madsen L. Building Emotional Awareness and Mental Health (BEAM): an open-pilot and feasibility study of a digital mental health and parenting intervention for mothers of infants. Pilot Feasibility Stud. 2023 Feb 18;9(1):27. doi: 10.1186/s40814-023-01245-x. PMID 36800982
- [Derived] MacKinnon AL, Simpson KM, Salisbury MR, Bobula J, Penner-Goeke L, Berard L, Rioux C, Giesbrecht GF, Giuliano R, Lebel C, Protudjer JLP, Reynolds K, Sauer-Zavala S, Soderstrom M, Tomfohr-Madsen LM, Roos LE. Building Emotional Awareness and Mental Health (BEAM): A Pilot Randomized Controlled Trial of an App-Based Program for Mothers of Toddlers. Front Psychiatry. 2022 Jun 24;13:880972. doi: 10.3389/fpsyt.2022.880972. eCollection 2022. PMID 35815022